CLINICAL TRIAL: NCT05078905
Title: Longitudinal Observations of Vaccine Responses to SARS-CoV-2 and Other Emerging Infectious Diseases
Brief Title: Vaccine Responses to SARS-CoV-2 and Other Emerging Infectious Diseases
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000688; 000688-I
Record Dates: First submitted 2021-10-13; First posted 2021-10-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01-20

CONDITIONS: COVID-19; Vaccination; Healthy Volunteer
Keywords: Vaccination; Pandemic; COVID-19; Pathogens; Immune Response; Natural History
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals Receiving Vaccine: Individuals receiving a vaccination for an emerging infection, like SARS-CoV-2

SUMMARY:
Background:

Vaccines against SARS-CoV-2, the virus that causes COVID-19, have been highly effective against preventing severe disease. But the protective effects of these vaccines appear to wane over time. Researchers want to learn why.

Objective:

To learn more about how the immune system responds to vaccines against infections like SARS-CoV-2.

Eligibility:

Healthy adults ages 18 or older who are scheduled to receive either a new vaccine or a booster shot against SARS-COV-2 or another emerging infection.

Design:

Participants will be screened with a medical history and blood and urine tests.

Participants will have up to 8 study visits in 1 year. Each visit should last less than 2 hours. At each visit, participants will give blood samples. Some blood samples will be used for genetic testing. They will also give updates on their health.

After the first study visit, participants will receive either a first vaccination or a booster shot. They must get the vaccine in their community or workplace. They will not get the vaccine at NIH.

This study currently focuses on SARS-CoV-2, but it will expand to other infectious diseases as they emerge and become the target of new vaccines.

...

DETAILED DESCRIPTION:
Study Description: This protocol will enroll up to 200 adults per year who are scheduled to be vaccinated against severe acute respiratory syndromecorona virus 2 (SARS-CoV-2) or other emerging pathogens. Participants will provide blood samples prior to and serially aftervaccination. The blood will be used to perform research studies of the immune response to primary (new) and secondary (booster) vaccines.

Objectives:

Primary Objective: Characterize longitudinal serologic and cellular responses to vaccination to SARS-CoV-2 and other emerging infections.

Secondary Objectives:

1. Evaluate baseline correlates of immune response to vaccination.
2. Correlate cellular and serologic responses after vaccination.
3. For vaccines that require two or more doses; characterize the immunologic responses following both the primary (new) and the secondary (booster) dose(s).
4. Evaluate the longevity of immune responses to primary (new) and secondary (booster) vaccination.

Endpoints: Primary Endpoint: Establish immunologically well characterized cohorts of primary (new) and secondary (booster) vaccinated individuals.

Secondary Endpoints: Establish factors associated with longevity of serologic and cellular responses to primary (new) and secondary (booster) vaccination.

ELIGIBILITY:
* INCLUSION CRITERIA:

General Inclusion Criteria for All Groups:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Age 18 years or older
3. Hemoglobin >= 9.0 grams per deciliter (g/dL) or >= 11.2 for women who are pregnant.
4. Willingness to give consent for the storage of blood samples for research
5. Ability of subject to understand and the willingness to sign a written informed consent document

Inclusion Criteria for Primary (New) Vaccination Group:

1. No history of having received a dose of the vaccine for the infectious disease being studied. Subjects who have enrolled under another Laboratory of Immunoregulation (LIR) protocol and had samples drawn prior to vaccination will also be eligible for enrollment.

Inclusion Criteria for Secondary (Booster) Vaccination Group:

1. Willingness to return for baseline research blood collection prior to booster vaccination.

EXCLUSION CRITERIA:

1. Current abuse of alcohol or other drugs that, in the judgement of the Principal Investigator (PI) could interfere with patient compliance.
2. Any medical or mental health condition that, in the judgement of the PI, would make the volunteer unable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals greater than 18 years of age who are scheduled to receive a initial or booster vaccination to an emerging infectious disease.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2050-01-01 (Estimated); Study Completion 2050-01-01 (Estimated)

PRIMARY OUTCOMES:
Characterize longitudinal serologic and cellular responses to vaccination to SARS-CoV-2 and other emerging infections. | throughout
  Establish immunologically well characterized cohorts of primary and secondary vaccinated individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Moir, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Identified data in BTRIS (automatic for activities in the Clinical Center). De-identified or identified data with approved outside collaborators under appropriate agreements. This study will comply with the NIH Genomic Data Sharing Policy, which applies to all NIH-funded research that generates large-scale human or non-human genomic data, as well as the use of these data for subsequent research. Large-scale data include genome-wide association studies (GWAS), single nucleotide polymorphisms (SNP) arrays, and genome sequence, transcriptomic, epigenomic, and gene expression data. De-identified data may be shared in an NIH-funded or approved public repositories, including the Database of Genotypes and Phenotypes (dbGAP) or in NCBI Virus Portal for viral sequencing.
Supporting Information: Study Protocol
Time Frame: Shared scientific data should be made accessible as soon as possible, and no later than the time of an associated publication, or the end of the award/support period, whichever comes first. Genomic data will be shared following the guidelines of the Genomic Data Sharing Policy, when applicable.
Access Criteria: Identified data in BTRIS (automatic for activities in the Clinical Center and will be available for use following the BTRIS Policy for Data Sharing and Use). De-identified or identified data with approved outside collaborators under appropriate agreements. De-identified genomic data may be shared in an NIH-funded or approved public repositories, including the Database of Genotypes and Phenotypes (dbGAP) and the use of the data within will be governed by their policies.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000688-I.html